CLINICAL TRIAL: NCT00467519
Title: Safety and Immunogenicity of Tdap Vaccine Compared to DTaP Vaccine as Fifth Dose Booster in Children 4 to 6 Years of Age
Brief Title: Safety and Immunogenicity of Tdap Vaccine Compared to DTaP Vaccine in Children 4 to 6 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TD517
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Results first posted 2010-12-03 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-01

CONDITIONS: Tetanus; Diphtheria; Pertussis
Keywords: Tetanus; Diphtheria; Pertussis; ADACEL; DAPTACEL
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough | interventions — adacel; Tetanus Toxoid; Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): DAPTACEL primed participants
  Interventions: Biological: Tdap (Tetanus Toxoid Reduced Diphtheria Toxoid/Acellular Pertussis)
- Group 2 (Experimental): Pentacel primed participants
  Interventions: Biological: DTaP (Diphtheria & Tetanus Toxoids & Acellular Pertussis Adsorbed)

INTERVENTIONS:
Biological: Tdap (Tetanus Toxoid Reduced Diphtheria Toxoid/Acellular Pertussis) — 0.5 mL, IM
  Other Names: Adacel
  Arms: Group 1
Biological: DTaP (Diphtheria & Tetanus Toxoids & Acellular Pertussis Adsorbed) — 0.5 mL, IM
  Other Names: DAPTACEL in the US; TRIPACEL in Canada
  Arms: Group 2

SUMMARY:
Currently, there is no 5-component acellular pertussis vaccine licensed for the 5th dose in US children aged 4 to 6 years.This study is aimed at providing evidence of sero-protection, booster response and safety of this formulation as a 5th dose.

Primary Objective:

- To compare the immune responses of Tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis (Tdap) Vaccine to Diphtheria, tetanus and acellular pertussis (DTaP) vaccine (all antigens) when each is administered as a 5th dose and given concurrently, to children aged 4 to 6 years.

Secondary/Observational Objectives:

* To compare the immune responses for pertussis antigens of Tdap Vaccine to DTaP vaccine (for pertussis antigens) when each is administered as a 5th dose and given concurrently, to children aged 4 to 6 years.
* To present the long-term immunogenicity at 1-, 3-, and 5-years post-vaccination after each long-term follow-up.
* To describe the safety profile following vaccine administration.

ELIGIBILITY:
Inclusion Criteria :

* Healthy, as determined by medical history and physical examination.
* Aged 4 to 6 (< 7) years at the time of study vaccination on Day 0.
* Signed and dated informed consent form that has been approved by the Institutional Review Board (IRB) by the parent or legally authorized representative.
* Signed and dated informed assent form from the subject if required by the IRB.
* Able to attend scheduled visits at Visit 1 and Visit 2 and able to comply with all trial procedures. Subjects will be invited to participate in the long-term immunogenicity follow-up study but a commitment to participate in the long-term is not required as an inclusion criterion.
* Documented vaccination history of 4 previous doses of DAPTACEL according to the recommended national immunization schedule for Diphtheria, tetanus and acellular pertussis (DTaP).

Exclusion Criteria :

* Participation in another clinical trial in the 4 weeks preceding the trial vaccination.
* Planned participation in another clinical trial during the original trial period.
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* Systemic hypersensitivity to any of the vaccine components or history of life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Blood or blood-derived products received in the past 3 months.
* Receipt of any other vaccine within 30 days prior to study vaccination, or planning to receive another vaccine within 30 days before the Visit 2 blood draw (with the exception of the annual influenza vaccine).
* History of diphtheria, tetanus or pertussis infection (confirmed either serologically or microbiologically).
* Thrombocytopenia or bleeding disorder contraindicating intra muscular vaccination.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1045 (Actual)
Dates: Start 2007-04; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (38):
- United States (37):
  - Birmingham, Alabama
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Fountain Valley, California
  - Huntington Beach, California
  - Oakland, California
  - Roseville, California
  - Sacramento, California
  - Norwich, Connecticut
  - Marietta, Georgia
  - Woodstock, Georgia
  - Bardstown, Kentucky
  - Crestview Hills, Kentucky
  - Louisville, Kentucky
  - Bossier City, Louisiana
  - Frederick, Maryland
  - Bellevue, Nebraska
  - Omaha, Nebraska
  - Rochester, New York
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Gresham, Oregon
  - Erie, Pennsylvania
  - Norristown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Rydal, Pennsylvania
  - Uniontown, Pennsylvania
  - Kingsport, Tennessee
  - Tullahoma, Tennessee
  - San Antonio, Texas
  - Layton, Utah
  - Springville, Utah
  - Chesapeake, Virginia
  - Midlothian, Virginia
  - Spokane, Washington
  - La Crosse, Wisconsin
- Edmonton, Alberta, Canada

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 13 April 2007 to 16 October 2009 in 42 clinical centers in the US and 1 clinical center in Canada.
Pre-assignment Details: A total of 1042 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Tdap Vaccine Group: Participants 4 to 6 years of age who had previously received 4 doses of Pentacel or DAPTACEL received a booster dose of tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed (Tdap).
- DTaP Vaccine Group: Participants 4 to 6 years of age who had previously received 4 doses of Pentacel or DAPTACEL received a booster dose of diphtheria, tetanus and acellular pertussis vaccine (DTaP).
Period: Overall Study
Arm/Group | Tdap Vaccine Group | DTaP Vaccine Group
Started | 531 | 511
Completed | 517 | 488
Not Completed | 14 | 23
Not completed — Protocol Violation | 8 | 4
Not completed — Lost to Follow-up | 2 | 9
Not completed — Withdrawal by Subject | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tdap Vaccine Group | DTaP Vaccine Group | Total
Number analyzed (Participants) | 531 | 511 | 1042
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 531 | 511 | 1042
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.45 (0.48) | 4.42 (0.47) | 4.44 (0.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 244 | 519
  Male | 256 | 267 | 523
Region of Enrollment [Number; unit: participants]
  United States | 522 | 502 | 1024
  Canada | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Seroprotection at Baseline and 30 Days Post-vaccination for Diphtheria and Tetanus at ≥ 0.1 IU/mL Level
Description: Seroprotection rate at level ≥ 0.1 IU/mL was defined as antibody concentrations ≥ 0.1 IU/mL.
  Diphtheria titers were determined by toxin neutralization assay; tetanus titers were determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Pre-dose and 30 days post-vaccination
Population: Diphtheria and tetanus antibody analysis was in all enrolled and vaccinated participants in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tdap Vaccine Group | DTaP Vaccine Group
Number analyzed (Participants) | 442 | 426
Percentage of Participants
  Diphtheria (IU/mL), Pre-dose [n = 442, 425] | 65 | 69
  Diphtheria (IU/mL), Post-dose [n = 442, 426] | 100 | 100
  Tetanus (IU/mL), Pre-dose [n = 442, 426] | 81 | 85
  Tetanus (IU/mL), Post-dose [n = 442, 426] | 100 | 100

2. Primary Outcome: Percentage of Participants Who Achieved Serothreshold at Baseline and 30 Days Post-vaccination for Diphtheria and Tetanus at Level ≥ 1.0 IU/mL
Description: Serothreshold rate at level ≥ 1.0 IU/mL was defined as antibody concentrations ≥ 1.0 IU/mL.
  Diphtheria titers were determined by toxin neutralization assay; tetanus titers were determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Pre-dose and 30 days post-vaccination
Population: Diphtheria and tetanus antibody analysis was in all enrolled and vaccinated participants in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tdap Vaccine Group | DTaP Vaccine Group
Number analyzed (Participants) | 442 | 426
Percentage of Participants
  Diphtheria (IU/mL), Pre-dose | 4 | 7
  Diphtheria (IU/mL), Post-dose | 99 | 100
  Tetanus (IU/mL), Pre-dose | 11 | 12
  Tetanus (IU/mL), Post-dose | 97 | 98

3. Primary Outcome: Percentage of Participants Who Demonstrated Booster Response at 30 Days Post-Vaccination for Pertussis
Description: Booster response was defined as post titer ≥ 0.4 IU/mL and pre-titer < 0.1 IU/mL, or Post/Pre titer ≥ 4 increase and pre titer ≥ 0.1 IU/mL but < 2 IU/mL, or Post/Pre titer ≥ 2 increase and pre-titer ≥ 2 IU/mL
  Post-vaccination titers for pertussis toxoid (PT), pertussis filamentous hemagglutinin (FHA), pertussis pertactin (PRN), and pertussis Fimbriae types 2 and 3 (FIM), were determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: 30 Days post-vaccination
Population: Pertussis antibody booster response analysis was in all enrolled and vaccinated participants in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tdap Vaccine Group | DTaP Vaccine Group
Number analyzed (Participants) | 441 | 423
Percentage of Participants
  Pertussis Toxoid (EU/mL) [n = 401, 387] | 88 | 94
  Filamentous Haemagglutinin (EU/mL) [n = 432, 407] | 92 | 89
  Pertactin (EU/mL) [n = 441, 423] | 92 | 95
  Fimbriae types 2 and 3 (EU/mL) [n = 432, 418] | 95 | 94

4. Other Pre Specified Outcome: Number of Participants Reporting at Least 1 Solicited Injection Site or Solicited Systemic Reaction Post-vaccination
Description: Solicited Injection Site Reactions: Pain, erythema/redness, swelling, increased left limb circumference, and increased right limb circumference. Solicited Systemic Reactions: Fever (temperature), headache, malaise, and myalgia.
Time Frame: Days 0 to 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Tdap Vaccine Group | DTaP Vaccine Group
Number analyzed (Participants) | 531 | 511
Participants
  Any Solicited Injection Site Reaction [n=529, 495] | 455 | 451
  Any Pain [n = 529, 495] | 318 | 334
  Grade 3 Pain (Incapacitating) | 1 | 4
  Any Erythema [n = 529, 494] | 140 | 201
  Grade 3 Erythema (> 50 mm) | 17 | 65
  Any Swelling [n = 529, 493] | 100 | 144
  Grade 3 Swelling (> 50 mm) | 8 | 23
  Any Increased Left Limb Circumference [n=527, 494] | 309 | 353
  Grade 3 Left Limb Circumference (> 40 mm increase) | 1 | 5
  Any Increased Right Limb Circumference [n=527, 494 | 241 | 244
  Grade 3 Right Limb Circumerence (> 40 mm increase) | 1 | 0
  Any Solicited System Reaction [n = 529, 495] | 256 | 260
  Any Fever [n = 527, 493] | 25 | 26
  Grade 3 Fever (> 39.5 °C) | 1 | 1
  Any Headache [n = 529, 495] | 60 | 74
  Grade 3 Headache (Prevents daily activities) | 3 | 4
  Any Malaise [n = 529, 495] | 143 | 150
  Grade 3 Malaise (Prevents daily activities) | 5 | 7
  Any Myalgia [n = 529, 495] | 185 | 196
  Grade 3 Myalgia (Prevents daily activities) | 3 | 8

5. Primary Outcome: Percentage of Participants Who Demonstrated Booster Response at 30 Days Post-Vaccination for Diphtheria and Tetanus
Description: Booster response was defined as post titer ≥ 0.4 IU/mL and pre titer < 0.1 IU/mL, or Post/Pre titer ≥ 4 increase and pre-titer ≥ 0.1 IU/mL but < 2 IU/mL, or Post/Pre titer ≥ 2 increase and pre-titer ≥ 2 IU/mL.
  Post-vaccination titers for Diphtheria was determined by neutralization assay; tetanus titers was determined by an enzyme-linked immunosorbent assay (ELISA).
Time Frame: 30 Days post-vaccination
Population: Diphtheria and tetanus antibody booster response were analysed in all enrolled and vaccinated participants, per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tdap Vaccine Group | DTaP Vaccine Group
Number analyzed (Participants) | 442 | 426
Percentage of Participants
  Diphtheria (IU/mL) [n = 442, 425] | 99 | 99
  Tetanus (IU/mL) [n = 442, 426] | 98 | 97

6. Primary Outcome: Geometric Mean Titers (GMTs) at Baseline and 30 Days Post Vaccination for Pertussis
Description: Pre- and post-vaccination GMTs and their 95% confidence intervals for pertussis toxoid (PT), pertussis filamentous hemagglutinin (FHA), pertussis pertactin (PRN), and pertussis Fimbriae types 2 and 3 (FIM), were determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Pre-dose and 30 Days Post-vaccination
Population: Geometric mean titers were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Tdap Vaccine Group | DTaP Vaccine Group
Number analyzed (Participants) | 442 | 426
EU/mL
  Pertussis Toxoid, Pre-dose [n = 411, 390] | 4.58 [4.16 to 5.05] | 4.98 [4.49 to 5.51]
  Pertussis Toxoid, Post-dose [n = 430, 423] | 53.1 [49.3 to 57.2] | 86.4 [79.9 to 93.5]
  Filamentous Haemagglutinin, Pre-dose [n= 435, 408] | 7.56 [6.64 to 8.61] | 7.60 [6.59 to 8.76]
  Filamentous Haemagglutinin, Post-dose [n=439, 424] | 102 [93.1 to 111] | 86.5 [78.3 to 95.5]
  Pertactin, Pre-dose [n = 442, 424] | 9.31 [8.40 to 10.3] | 11.1 [10.0 to 12.4]
  Pertactin, Post-dose [n = 441, 425] | 121 [109 to 134] | 173 [155 to 193]
  Fimbriae types 2 and 3, Pre-dose [n = 434, 420] | 23.8 [21.0 to 27.0] | 24.4 [21.4 to 27.7]
  Fimbriae types 2 and 3, Post-dose [n = 439, 424] | 425 [387 to 467] | 388 [354 to 425]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the day of vaccination to 6 months post-vaccination.
Arm/Group | Tdap Vaccine Group | DTaP Vaccine Group
Serious Adverse Events (participants affected / at risk) | 4/531 | 5/511
Other Adverse Events (participants affected / at risk) | 318/531 | 353/511
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tdap Vaccine Group (N=531) | DTaP Vaccine Group (N=511)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Tdap Vaccine Group (N=531) | DTaP Vaccine Group (N=511)
Injection site Erythema (General disorders) | 140/529 (140) | 201/494 (201)
Fever (General disorders) | 25/527 (25) | 26/493 (26)
Increased left limb circumference (General disorders) | 309/527 (309) | 353/494 (353)
Increased right limb circumference (General disorders) | 241/527 (241) | 244/494 (244)
Injection site bruising (General disorders) | 28 (31) | 40 (42)
Injection site induration (General disorders) | 20 (21) | 28 (30)
Myalgia (Musculoskeletal and connective tissue disorders) | 185/529 (185) | 196/495 (196)
Headache (Nervous system disorders) | 60/529 (60) | 74/495 (74)
Cough (Respiratory, thoracic and mediastinal disorders) | 48 (49) | 29 (31)
Solicited Injection Site Pain (General disorders) | 318/529 (318) | 334/495 (334)
Solicited Injection Site Swelling (General disorders) | 100/529 (100) | 144/493 (144)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications